CLINICAL TRIAL: NCT03585088
Title: Can we Predict Postoperative Analgesic Requirement by Intraoperative Nociception?
Brief Title: The Prediction for Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC2018-04-129
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-05

CONDITIONS: Pain, Postoperative; Nociceptive Pain; Analgesia, Patient-Controlled; Analgesics
MeSH Terms: conditions — Pain, Postoperative; Nociceptive Pain; Agnosia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPI Group (Other): All patients who received the liver resection surgery will receive surgical pleth index
  Interventions: Device: surgical pleth index

INTERVENTIONS:
Device: surgical pleth index — All patients applied surgical pleth index after recovery of spontaneous breathing at the time of peritoneum and skin closure under Bispectral index score <=60.

SUMMARY:
If the individual patient's pain is assessed and the amount of analgesic needed after surgery is predicted, appropriate injection of pain control and excessive injection of narcotic analgesic can be prevented. Therefore, investigators try to evaluate the degree of pain during surgery and the amount of analgesic use for management of postoperative pain.

DETAILED DESCRIPTION:
Post-operative pain not only alleviates patient discomfort, but also delays recovery and thus prolongs the hospital stay. There are many ways to control postoperative pain, but analgesic infusion through venous route, patient controlled analgesia (PCA), especially narcotic analgesics, is often used to control the infusion when needed. However, because PCA is based on only age, weight, and underlying diseases, there are limitations in effective analgesia, and excessive sedation due to excessive infusion. Therefore, if the individual patient's pain is assessed and the amount of analgesic needed after surgery is predicted, appropriate injection of pain control and excessive injection of narcotic analgesic can be prevented. The noxious stimuli during surgery may have a negative effect on the healing process and surgical outcome of the wound due to stress reaction and catabolism, secretion of pituitary hormone, activation of the sympathetic nervous system, and immunological changes. Therefore, proper analgesia is needed during general anesthesia. A non-invasive, non-invasive analgesic device is currently available for Surgical pleth index (SPI) to assess the status of intraoperative analgesia. SPI = 100- (0.3 * heart beat interval + 0.7 * photoplethysmographic pulse wave amplitude) is automatically and continuously calculated from the waveform of peripheral oxygen saturation.

In the postoperative pain prediction study with SPI, the SPI value at the end of the operation was found to be proportional to the pain in the recovery room. However, only the pain score immediately after the operation was confirmed in these studies. Therefore, investigators try to evaluate the degree of pain during surgery and the amount of analgesic use for management of postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

undergoing liver resection (laparoscopic or laparotomy)

Exclusion Criteria:

patients who refused to participate patients who have cardiac arrythmia patients who have allergic history for remifentanil

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
The correlation of requirement of postoperative analgesics for postoperative 24 hours and intraoperative nociception score | intraoperative nociception score: 3 minutes during closure peritoneum and skin; requirement of postoperative analgesics: the first 24 hour in postoperative phase
  The consumption of patient controlled analgesia and intraoperative surgical pleth index score

SECONDARY OUTCOMES:
The correlation of requirement of postoperative analgesics for postoperative 6 hours and intraoperative nociception score | intraoperative nociception score: 3 minutes during closure peritoneum and skin; requirement of postoperative analgesics: the first 6 hour in postoperative phase
  The consumption of patient controlled analgesia and intraoperative surgical pleth index score
The correlation of requirement of postoperative analgesics for postoperative 48 hours and intraoperative nociception score | intraoperative nociception score: 3 minutes during closure peritoneum and skin; requirement of postoperative analgesics: the first 48 hour in postoperative phase
  The consumption of patient controlled analgesia and intraoperative surgical pleth index score
The correlation of postoperative pain score and intraoperative nociception score | awaken after general anesthesia in post-anesthesia care unit , postoperative 6, 24, 48 hours
  The postoperative pain score (numeric rating pain score, no pain=0~ worst pain=10)and intraoperative surgical pleth index score
The side effects of analgesics | awaken after general anesthesia in post-anesthesia care unit , postoperative 6, 24, 48 hours
  nausea/vomiting, sedation, itching, respiratory depression

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dolin SJ, Cashman JN. Tolerability of acute postoperative pain management: nausea, vomiting, sedation, pruritus, and urinary retention. Evidence from published data. Br J Anaesth. 2005 Nov;95(5):584-91. doi: 10.1093/bja/aei227. Epub 2005 Sep 16. PMID 16169893
- [Background] Ledowski T, Sommerfield D, Slevin L, Conrad J, von Ungern-Sternberg BS. Surgical pleth index: prediction of postoperative pain in children? Br J Anaesth. 2017 Nov 1;119(5):979-983. doi: 10.1093/bja/aex300. PMID 29028932
- [Background] Ledowski T, Burke J, Hruby J. Surgical pleth index: prediction of postoperative pain and influence of arousal. Br J Anaesth. 2016 Sep;117(3):371-4. doi: 10.1093/bja/aew226. PMID 27543532